CLINICAL TRIAL: NCT03206736
Title: The Effect of Loop Duodenal Switch Surgery in Morbidly Obese Patients on Weight Los at One Year.
Brief Title: Loop Duodenal Switch: Outcomes at One Year
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low study enrollment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0281-17-FB
Record Dates: First submitted 2017-06-22; First posted 2017-07-02 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Loop DS Patients (Experimental): Patients who receive a Loop DS procedure
  Interventions: Other: Loop DS surgery

INTERVENTIONS:
Other: Loop DS surgery — these patients will receive a loop DS bariatric procedure

SUMMARY:
The biliopancreatic diversion and duodenal switch (BPD-DS) is an accepted and published type of bariatric surgery in the United States. The BPD-DS procedure produces the most weight loss of any bariatric surgery commonly performed but has the highest risk of malnutrition and gastrointestinal side effects. The loop duodenal switch (L-DS) is a bariatric surgery which has been modified from a biliopancreatic diversion and duodenal switch to maintain excellent weight loss while possibly reducing side effects. The surgical modifications in this procedure include reducing the number of intestinal reconnections from two to one and reducing the amount of small intestine which is bypassed. The L-DS operation is considered experimental by the American Society of Metabolic and Bariatric Surgery as long-term data in large numbers of patients is not available for weight loss or side effects. The purpose of this study is to examine weight loss and other outcomes in the L-DS operation up to 1 year after the procedure.

Study participants will be seen in the clinic at 2 and 6 weeks, and 3, 6, 9, and 12 months per the bariatric surgery center protocol. As part of these normally scheduled visits, weight loss and health status will be recorded. Labs will be checked at 3, 6, and 12 months for nutritional status. A survey to reassess health-related quality of life and gastrointestinal symptoms will be performed at 3 months, 6 months and 12 months.

DETAILED DESCRIPTION:
1. Screening and Informed Consent Subjects will be screened on a weekly basis for eligibility of enrollment. If eligible, patients will be approached by study staff at the initial surgical consultation. The purpose of the study and risks of the procedures will be explained to the subject and the consent process must be documented accordingly in the medical record. Subjects who agree to study participation must sign an IRB approved informed consent form. Subjects will be informed that their participation in this study is voluntary and they may refuse to participate or discontinue from the study at any time. Subjects will be given the opportunity to ask the investigator questions so that they are adequately informed about the research. A copy of the signed informed consent must be provided to the subject and the informed consent process will be documented in source documents. If new information becomes available that may affect a subject's decision to continue to take part in the study, this information will be discussed with the subject by the investigator.

Failure to meet submission requirements:

Each patient will be required to meet their individual insurance companies requirements for submission of bariatric surgery approval. Subjects who provide study consent but then do not submit for insurance approval or are denied will be considered "discontinued" and will not require additional study follow-up visits. The reason for the discontinuation will be clearly delineated on the applicable case report form. Subjects in who the L-DS procedure is begun but not completed will be considered "discontinued" once discharged from the hospital and not require any additional study follow-up visits. Reasons for discontinuation will be recorded in the case report form. Additionally, female patients of child bearing age will undergo a standard of care pregnancy test at the time of the pre-operative surgical testing (2/3 weeks before surgery) and always the morning of surgery by urine HCG.

Surgical Procedures:

The operation will be performed per standard of care and as previously described (1-3), with the exception that in this protocol the duodeno-intestinal anastomosis will be performed at approximately 300 cc with moderate stretch from the ileocecal valve, rather than 200 cm or 250 cm, as in previous reports. The purpose of this change is to allow greater nutrient absorption since a previous report observed no difference in mean excess weight loss between 200 cm and 250 cm (Sanchez-Pernaute 2013). In addition, the sleeve gastrectomy will be performed over a 40 French bougie. The duodeno-intestinal anastomosis will be hand-sewn. Subjects will be maintained on a low-calorie diet for the first post-operative month, as per standard of care. In addition, multivitamin supplements, calcium, and iron should be prescribed and maintained per standard of care.

Schedule:

Subjects will be evaluated preoperatively, during the procedure, at discharge, and at 2 weeks, 6 weeks, 3 months, 6 months, 9 months, and 12 months. Assessments to be conducted/data collected at each visit are listed below and in the study assessments table.

1. Pre-operative Assessment The following assessments will be performed pre-operatively prior to the scheduled surgical procedure and the results recorded on the appropriate subject report form Verification of pre-operative eligibility criteria Subject demographics (gender, age, race, ethnicity, smoking history) Height, weight, and body mass index (BMI) Comorbidity assessment (prevalence and duration of type 2 diabetes mellitus, sleep apnea, hypertension, dyslipidemia/hyperlipidemia, and other clinically relevant comorbidities as determined by the treating physician), including medications Fasting labs (glucose, hemoglobin, HbA1C, hematocrit, ferritin, albumin, total protein, calcium, parathyroid hormone, vitamin A, Vitamin B1, Vitamin B12, Vitamin D2/3, Vitamin 3, Vitamin K, folic acid, insulin, lipid panel, triglycerides, total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), C-peptides, iron, copper, and zinc) Surgical history Health- related Quality of life, as measured by the SF-36 assessment Gastrointestinal symptom rating scale, as measured by the GSRS form GERD HR-QL Pre-operative Dietary Restrictions
2. Operative Assessment The following procedures and assessments will be performed on the day of/during the procedure: Weight and BMI American Society of Anesthesiologists (ASA) grade operative time (defined as skin to skin time) anesthesia start and stop time estimated blood loss adverse events surgical technique (eg protocol requires: 40 French bougie, distal gastrectomy starting 5 cm distal to the pylorus, duodeno-intestinal anastomosis performed at approximately 300 cm from the ileocecal valve, hand-sewn anastomosis, and fascia closure for all port sites accommodating trocars greater than 12 mm) surgical conversions to open concomitant procedures performed during the procedure
3. Discharge Assessment

   The following procedures and assessments will be performed prior to discharge:

   Length of hospital stay Surgical site infection assessment Surgical site infection (SSI) Adverse events (see below)
4. Post-operative follow-up assessments The following procedures and assessments will be performed at 2 weeks, 6 weeks, 3 months, 6 months, 9 months and 12 months post procedure (+/- 7 days for 2 and 6 week follow-up, +/- 14 day days for all other months).

   Post-operative standard of care:

   Compliance with prescribed dietary supplements Weight and BMI EWL Comorbidity assessment (prevalence and duration of type 2 diabetes mellitus, sleep apnea, hypertension, dyslipidemia/hyperlipidemia, and other clinically relevant comorbidities as determined by the treating physician), including medications and relevant lab tests per standard of care at 3, 6, and 12 months (glucose, hemoglobin, HbA1C, hematocrit, ferritin, albumin, total protein, calcium, parathyroid hormone, vitamin A, Vitamin B1, Vitamin B12, Vitamin D2/3, Vitamin 3, Vitamin K, folic acid, insulin, lipid panel, triglycerides, total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), C-peptides, iron, copper, and zinc) Surgical site infection assessment at 1 month only health-related quality of life (HR-QOL) (SF-36), GERD-HRQL and GSRS questionnaire expressed as change from baseline at 3, 6 and 12 months only need for endoscopy adverse events (see below)
5. Adverse Events Adverse events for all bariatric procedures are tracked within our centers Metabolic and Bariatric Surgery Accreditation and Quality Improvement Program (MBSAQIP) database. All bariatric centers accredited by the American Society for Metabolic and Bariatric Surgery (ASMBS) are required to submit all bariatric surgery data, including experimental procedures like the L-DS, to the MBSAQIP database for quality review. Our bariatric surgery team has open access to our centers data for quality review purposes and will compare adverse events for the L-DS to the other procedures performed by our center. Adverse events are categorized by organ system (wound, respiratory, urinary tract, CNS, cardiac, or other) as specified by the MBSAQIP. Any post-operative occurrence within 30 days will be documented if related to the bariatric procedure. Bariatric related readmission and reoperations are also tracked per MBSAQIP guidelines. The L-DS would be stopped if a statistically significant increase in morbidity, mortality, or failed weight loss is found compared to the centers other commonly performed bariatric procedures.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be 19-70 years of age at the time of enrollment.
2. The subject must be willing and able to participate in the study procedures and to understand and sign the informed consent.
3. The subject is under consideration for surgery for obesity or metabolic disease and elects to undergo a primary loop duodenal switch procedure or as a conversion procedure for failed, sustained weight loss after a sleeve gastrectomy or laparoscopic adjustable gastric band performed more than 12 months prior to time of evaluation.
4. The subject has a BMI of greater than or equal to 40 kg/m2 at time of surgical consultation.

Exclusion Criteria:

1. Subjects under 19 years of age or older than 70 years of age
2. Subject is not willing or able to participate in the study procedures and understand the informed consent.
3. The subject wishes to under a different bariatric procedure other than the loop duodenal switch.
4. The subject has a BMI of less than 40 kg/m2 at the time of surgical consultation.
5. Any female subject who is pregnant, or is actively breast-feeding
6. Any subject who is considered to be part of a vulnerable population (eg. prisoners or those with psychological concerns or those without sufficient mental capacity)
7. The procedure is an emergency procedure

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Excess weight loss | 1 year
  Excess weight loss at 1 year will be measured by comparing BMI at 1 year to the presurgical BMI. Body mass index (BMI) is calculated using the patient's height and weight. Height will be measured using a stadiometer and weight will be measured using the clinic's bariatric scale

SECONDARY OUTCOMES:
anesthesia | at surgery
  Anesthesia start and stop time
Blood loss | at surgery
  Estimated blood loss during surgery
Surgery conversion | at surgery
  surgical conversions to open procedure
Concomitant procedures | at surgery
  Concomitant procedures performed during the procedure
Hospital LOS | at surgery
  Length of hospital stay for the surgical procedure
Surgical site infection | 1 year
  Development of a surgical site infection.
T2DM | 1 year
  Prevalence and duration of type 2 diabetes mellitus
Sleep apnea | 1 year
  Sleep apnea
Hypertension | 1 year
  Hypertension
Lipids | 1 year
  dyslipidemia/hyperlipidemia
changes in quality of life | 1 year
  Patient quality of life will be assessed using an SF-36 questionnaire administered prior to the surgery and at 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Kothari, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data with other researchers.